CLINICAL TRIAL: NCT05169359
Title: Empowering Veterans to Actively Communicate and Engage in Shared Decision Making in Medical Visits, A Randomized Controlled Trial
Acronym: ACTIVet-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 19-442
Record Dates: First submitted 2021-12-02; First posted 2021-12-23 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus (Type 2)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Stepped wedge design
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Other): The study is a type 2 hybrid Effectiveness Implementation trial. The study uses a stepped wedge design. Patients are in a usual care phase until their clinic begins active implementation. Once active implementation begins, patients will view the Speak Up! Video intervention prior to their visit. The 10-minute video program will be provided to patients for viewing on an iPad (or other modality such as a portable DVD player, computer, or TV as appropriate to the site based on PDSA activities during implementation planning). Nurses may also send a video link to the patient via secured messaging as a method of watching the video before the primary care visit.
  Interventions: Behavioral: Speak Up! Video

INTERVENTIONS:
Behavioral: Speak Up! Video — Once a clinic begins active implementation (is ready to show the video) patients will view the Speak Up! Video intervention prior to their visit. The 10-minute video program will be provided to patients for viewing on an iPad (or a portable DVD player, computer or TV as appropriate to the site based on PDSA activities during implementation planning). The clinic staff will set patients up with comfortable headphones.

SUMMARY:
Type 2 diabetes is a significant condition in VA affecting 20% of VA patients. Adherence to medication regimens and lifestyle factors is important to achieve care goals for these patients. Patients who use active participatory communication behaviors with their providers have better adherence to treatment and better biomedical outcomes, yet many patients are not prepared to engage in active communication with their providers. Existing coaching interventions have not been adopted in practice because of the cost of trained personnel. The investigators have shown the efficacy of a low-cost video that did not require trained personnel. This proposal proposes to test implementation strategies to deliver that video in VA primary care clinics and to test the effectiveness of the video to improve outcomes in a Hybrid Type 2 effectiveness-implementation trial using a cluster randomized stepped wedge design at eight sites. This proposal will test feasibility of implementing the video and if successful will generate the evidence to justify widespread dissemination of the video.

DETAILED DESCRIPTION:
Background: Type 2 diabetes mellitus (T2D) affects almost one in five VA patients overall and almost one in four VA patients who are racial and ethnic minorities. Adherence to medication regimens and lifestyle factors (such as diet and exercise) is important to improve outcomes in T2D. Adherence to these factors and subsequent achievement of outcomes is related, at least in part, to effective communication in medical encounters. Empowering and activating patients to use more effective communication behaviors with their providers leads to better adherence to treatment and better biomedical outcomes. However, interventions to improve communication have not been adopted in practice largely due to the cost of trained personnel to deliver the training. Thus, there is a gap in effective interventions that can improve communication related outcomes. In a recent VA HSR&D funded trial the investigators showed efficacy of the Speak Up! video. Veterans watching the video had significantly higher self-efficacy to communicate and lower hemoglobin A1c at follow-up.

Significance: Type 2 diabetes (T2D) is common, expensive, and chronic. Estimates put the prevalence of T2D at almost 20 percent. The proposed study is highly significant because the condition under study, T2D, is highly prevalent and has negative impacts for Veterans with the symptoms and sequelae of T2D. The objective to activate patients' communication to achieve goals of care and to improve outcomes of T2D is responsive to VA priorities to improve customer service, primary care practice, and care of complex chronic diseases.

Innovation: The proposal to engage patients in communication in medical visits is innovative because addressing patients' communication as contrasted with providers' communication is unique in the VA. It is also innovative because activating patients facilitates patient-centered care and shared decision making which are key goals in the VA/DOD guideline for the management of T2D and contributes to VA's commitment to the Whole Health model. Also, the intervention could be a paradigm for encouraging patients with other conditions to use active participatory communication. Specifically, the design and communication content of Speak Up! Could serve as a model for the development of activation interventions for Veterans with other conditions.

Specific Aims: The proposed Hybrid Type 2 study has two specific aims:

Aim 1. Implementation aim - In partnership with key clinical staff develop a strategy to deliver the Speak Up! video in VA outpatient primary care clinics using a facilitated Plan Do Study Act (PDSA) process.

Aim 2. Effectiveness aim - Examine the effectiveness of the Speak Up! video using the RE-AIM framework to evaluate Reach into the patient population, Effectiveness to improve outcomes (Hemoglobin A1c, communication self-efficacy, diabetes distress), Adoption by providers and clinics, Implementation (completion, fidelity, and intensity), and Maintenance after the end of external facilitation.

Hypothesis 1. Patients will have improvements in outcomes (A1c, diabetes distress, communication self-efficacy) from before to after watching the video.

Exploratory Hypothesis 2. Patients that are at higher risk of having challenges communicating with physicians (patients with low health literacy, African-American patients, patients with depression) will also have improvements in outcomes.

Methodology: The proposed study is a Hybrid Type 2 effectiveness - implementation trial of the intervention using a cluster-randomized stepped-wedge design in eight clinics. The investigators will test the implementation strategies using a formative evaluation guided by the Promoting Action on Research Implementation in Health Services (PARIHS) framework, and the investigators will use the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework: to examine effectiveness of the Speak Up! Video; to supplement the formative evaluation from PARIHS; and to conduct a summative evaluation to evaluate success of the implementation strategies.

Implementation/Next Steps: This proposal will test the feasibility of implementing the Speak Up! video in primary care and if successful will generate the evidence to justify widespread dissemination of the video.

ELIGIBILITY:
Inclusion Criteria:

* Dx of T2D
* Hemoglobin A1c ("A1c") 7 or greater
* Adults, age 18 or older
* Visit at a participating site
* Receives care from primary care provider more than once a year at VA

Exclusion Criteria:

* Lives in skilled nursing facility
* Dementia (abnormal SBT)63
* Creatinine >3 (or eGFR<20), recent MI or admission for HF
* Terminal medical condition
* Drug- (e.g., steroid) induced diabetes.
* Blind or deaf (e.g., unable to view/hear video

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HgbA1c at 3 months post-visit | Collected at baseline and 3 months post-visit
  HgbA1c is regarded as the standard laboratory measurement (blood test) for assessing the control of diabetes over approximately three months preceding the test. HgbA1c is usually checked several times a year in patients with poorly controlled diabetes.
Change from pre-visit communication self-efficacy score at 1 week post visit | Collected at pre-visit and 1 week post-visit
  Communication Self-Efficacy (pre and post visit) is the degree to which a patient feels able to interact with his/her provider in order to provide information about problems, obtain desired information about diagnosis, treatment and prognosis, and participate in formulating a plan. The Perceived Efficacy in Physician-Patient Interactions scale (PEPPI) is a valid and reliable measure of patients' perceived self-efficacy in interacting with physicians (alpha 0.83). The short form of the PEPPI (PEPPI-5) has 5-items. Score on the PEPPI-5 ranges from 5-25. Higher scores reflect a better perceived self-efficacy in interacting with physicians.
Change from pre-visit diabetes distress score at 1 week post visit | Collected at pre-visit and 1 week post-visit
  Diabetes Distress is a 17-item scale that measures the emotional burden of diabetes on four subscales: emotional burden, physician-related distress, regimen-related distress, and diabetes-related interpersonal distress subscale. The Diabetes Distress scale is internally consistent and is well correlated with measures of depression, meal planning, exercise, and cholesterol levels. The scale ranges from 17 to 102. Higher scores indicate higher distress.

SECONDARY OUTCOMES:
Change from baseline trust in provider score at 1 week post visit | Collected at baseline and 1 week post-visit
  Trust in Provider is measured pre- and post visit using a 5-item measure. The scale is scored on a 7-point Likert scale using the anchors "strongly disagree" and "strongly agree". The scale ranges from 5 to 35. Higher scores reflect higher trust in provider.
Change from pre-visit patient engagement score at 1 week post visit | Collected at pre-visit and 1 week post-visit
  Patient Engagement is assessed with the Altarum Consumer Engagement (ACE) measure. We use 8-items from two subscales (commitment and navigation). The scale ranges from 8 to 40. Higher scores are associated with higher patient's engagement in their healthcare.
Change from pre-visit medication adherence at 1 week post visit | Collected at pre-visit and 1 week post-visit
  This measure of medication adherence is the 9-item Brief Medication Questionnaire (BMQ), a highly sensitive scale for identifying non-adherence. The scale ranges from 9 to 45. Higher scores indicate more non-adherence.
Change from pre-visit self-care score at 1 week post visit | Collected at pre-visit and 1 week post-visit
  Self-Care will be measured with the Summary of Diabetes Self Care Activities (SDSCA) a well validated measure that assesses self-care activities (e.g., diet, physical activity, and smoking) The scale ranges from 12 to 96. Higher scores indicate better diabetes self-care.
Shared decision making | Collected 1 week post visit
  Shared Decision Making (SDM) will be measured with the CollaboRATE. The scale ranges from 0 to 27. Higher scores indicate higher shared decision making. This measure assesses discussion of options, pros, cons and preferences of a health decision. Higher scores indicate greater shared decision making.
Communication Ratings | Collected 1 week post visit
  The questionnaire assesses patients' ratings of their own participatory communication behavior. It is a 5-item scale. The scale is scored from 1 (completely disagree) to 7 (completely agree). The higher scores indicate a better quality of communication. The scale ranges from 5 to 35.
Patient Centered Care | Collected 1 week post visit
  Patient-Centered Care is measured with the Consultation Care Measure (CCM). The CCM measures patients' ratings of their provider on five subscales. The scale ranges from 21 to 105. Higher scores are associated with higher patient ratings of their provider.
Change from pre-visit medication adherence at 3 months post visit | Collected at pre-visit and 3 months post visit
  Medication adherence will also be assessed with a medication possession ratio (MPR) for diabetes medications. MPR will be based on VA pharmacy data. MPR is a ratio of the number of days the patient has drug in their possession divided by the number of days in the follow-up period (MPR = days with drug / total days). The investigators will use a mean MPR for patients on multiple oral hypoglycemic medications.
Change from baseline functional status score at 1 week post visit | Collected at baseline and 1 week post visit
  Functional Status will be assessed with the Veterans RAND-12 (VR-12), a patient-reported global-health measure of physical and mental health status and that has a non-proprietary scoring algorithm. The scale is normalized to a range from 0-100; higher scores indicate better functional status.
Change from pre-visit self-management score at 1 week post visit | Collected at pre-visit and 1 week post visit
  Diabetes self-management will be measured using the Diabetes Management Self Efficacy (DMSE) scale (alpha 0.91). This scale has 20 items. The scale ranges from 20 to 80. Higher scores indicate better diabetes self-management.
Promis | Change from baseline promis score at 1 week post visit
  Patient engagement will be assessed with the PROMIS Healthcare engagement measure including 8 items. Scores range from 8-40. Higher scores indicate higher healthcare engagement for patients.

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Gordon, MD BS, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (3):
- United States (3):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Adam Benjamin Jr VA Outpatient Clinic, Crown Point, IN, Crown Point, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Final datasets underlying all publications resulting from the proposed research will not be shared outside VA, except as required under the Freedom of Information Act (FOIA), for the for the following reasons: Data will be collected and accessed with a waiver of HIPAA authorization and as such disclosure outside the VA is restricted. For appropriate requests we will seek IRB and privacy officer approval for release of de-identified anonymized data.
Supporting Information: Study Protocol
URL: https://bcove.video/3jEBVS2

DOCUMENTS (1):
  • Informed Consent Form (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT05169359/ICF_000.pdf